CLINICAL TRIAL: NCT05917353
Title: A Randomized Control Trial of Hinex Jelly on the Changes in Muscle Quality and Quantity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(I)-20220124
Record Dates: First submitted 2023-06-05; First posted 2023-06-23 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-06

CONDITIONS: Nutrition, Healthy; Muscle Weakness; Elderly
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hinex Jelly Nutritional Supplement Intervention Group (Experimental): Week 0th, Week 4th (14 days before and after), Week 8th (14 days before and after), Week 12th (14 days before and after), diet and exercise health education was given, with daily intervention of Hinex Jelly nutritional supplements 1 serving per day during 0th to 8th Week;
  Interventions: Dietary Supplement: Hinex Jelly
- Routine care group (No Intervention): Week 0th, Week 4th (14 days before and after), Week 8th (14 days before and after), Week 12th (14 days before and after), the subjects were given regular dietary and exercise health education.

INTERVENTIONS:
Dietary Supplement: Hinex Jelly — 1. Name: Hinex Jelly
  2. Dosage form: Semi-solid jelly/ A-114001297-00000-2
  3. Dose(s): 300g/pack (per serving)
  4. Dosing schedule: one pack (serving) per day
  5. Mechanism of action: Nutritional supplement semi-solid food (content 61-91g/100g, protein 4.0-6.0/100g, saturated fatty acid 0.72-1.08g/100g, carbohydrate 12.56-18.84g/100g, dietary fiber 1.0-1.4g/100g), It is used as a nutritional supplement food.
  Arms: Hinex Jelly Nutritional Supplement Intervention Group

SUMMARY:
Taiwan is about to enter a super-aged society in 2025. The health problems of the elderly are getting more and more attention. Among these geriatric issues, sarcopenia is an important issue. Sarcopenia is the culprit of disability in old age. It is characterized by persistent and general loss of skeletal muscle mass and function throughout the body, which may lead to disability, decreased quality of life, and even inability to take care of yourself and an increased risk of death. Human skeletal muscle decreases with age. After the age of 40, muscle mass will be lost at a rate of 8% per decade; after the age of 70, it will be lost at a faster rate of 15% per decade in average. Although all elderly will lose muscle mass due to aging, the degree and speed of loss vary from person to person. In addition to aging, it may also be caused by chronic diseases.

Exercise intervention and nutritional intervention are the first choices for sarcopenia intervention. Regarding nutritional requirements, the elderly need at least 15 grams of essential amino acids per day for muscle building. Among them, leucine is the most important, which can increase protein production and reduce decomposition. Foods rich in leucine include soybeans, fish or beef. However, elderly people may not be able to get enough protein from their daily diet smoothly, often because of dysphagia, such as dental problems or chewing and swallowing problems. Therefore, oral nutritional supplements are relatively important for the improvement of muscle mass. Nutritional Supplement Hinex Jelly has 303 calories per serving, contains up to 15g of high-quality protein and a high amount of branched-chain amino acids, which is beneficial for muscle synthesis and tissue repair, plus a variety of minerals, vitamins, water-soluble dietary fiber, hydrolyzed collagen and other ingredients can strengthen nutritional supplements, maintain good health.

In summary, this study intends to explore the effect of Hinex Jelly nutritional supplemental intervention on muscle mass quality and quantity changes by means of randomized intervention and controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 50 (include 50 years old).
* Can cooperate with the study.
* No surgical intervention within 3 months.

Exclusion Criteria:

* Those who have obvious difficulty in movement (such as amputation) and cannot cooperate with the study.
* Those who are equipped with pacemakers or internal electronic medical devices.
* Pregnant women.
* Use of drugs or interventional therapy that may affect changes in body weight or muscle mass (such as other oral nutritional supplements, medicine, weight reduction medicine, bariatric gastric endoscopy therapy, bariatric surgery, acupuncture, acupuncture, electrical stimulation, etc.).
* Allergic to dairy or soy products.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Appendicular skeletal muscle mass index at 8 weeks | 8 weeks after the first session
  Appendicular skeletal muscle mass index assessed using the Inbody S10
Change from Baseline handgrip strength at 8 weeks | 8 weeks after the first session
  assessed with a Jamar handheld dynamometer in kilograms
Change from Baseline performance on the 5-repetition sit-to-stand test at 8 weeks | 8 weeks after the first session
  assessed in seconds
Change from Baseline performance on 6-metre walk test at 8 weeks | 8 weeks after the first session
  assessed in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No